CLINICAL TRIAL: NCT00070681
Title: Outcomes of Sleep Disorders in Older Men
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 158; R01HL070848 (NIH)
Record Dates: First submitted 2003-10-06; First posted 2003-10-09 (Estimated); Last update posted 2016-07-29 (Estimated); Status verified 2009-04

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Sleep; Sleep Apnea Syndromes; Neurologic Manifestations; Osteoporosis; Bone Diseases
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Sleep Apnea Syndromes; Neurologic Manifestations; Osteoporosis; Bone Diseases

INTERVENTIONS:
Procedure: Polysomnography

SUMMARY:
To determine the effects of sleep disorders on cardiovascular function and disease in older men.

DETAILED DESCRIPTION:
BACKGROUND:

It is estimated that over 50 percent of adults aged 65 and older report some sleep disruption, while about 20 percent suffer from chronic insomnia. Obstructive sleep apnea, a major cause of daytime drowsiness, occurs in an estimated 20-60 percent of older people, depending on the definition used and the specific population being studied. Despite the high prevalence of sleep disorders in the elderly, there have been relatively few studies focused on the consequences. Most studies have been limited by cross-sectional design, small sample size, or lack of comprehensive and objective assessment of sleep. The study, Outcomes of Sleep Disorders in Older Men, will take advantage of the established cohort that has been recruited for the Osteoporotic Fractures in Men (MrOS) Study (5U01AR045647-Dr. Eric Orwoll, PI). MrOS, a 7-year study that began in July 1999, is a multi-center prospective study of approximately 6,000 men aged 65 and older. During the MrOS baseline visit, a broad variety of measurements were collected, including body composition and body fat distribution by dual energy X-ray absorptiometry (DEXA) and quantitative computed tomography, bone density, anthropometry, performance-based tests of strength and balance, medical history, medication use, smoking and alcohol use, and other parameters. Blood, urine, and DNA specimens have been archived for use in future studies of importance to the health of older men.

DESIGN NARRATIVE:

In a subcohort of 3,000 MrOS participants, comprehensive and accurate assessments of sleep will be added using in-home polysomnography, wrist actigraphy, questionnaires and other measures; and prospective adjudication of cardiovascular disease (CVD) events, to the extensive measures that have already been performed or planned in the MrOS cohort study. These new measures will enable testing of several important hypotheses: 1) to characterize the associations between sleep disruption and subsequent CVD events during 3.5 years of follow-up, 2) to determine if sleep disturbances are associated with an increased risk of total and cause-specific mortality in older men, 3) to test whether sleep disturbances are associated with increased risk of falls and decreased physical function, 4) to test whether sleep disturbances are associated with impaired cognitive function in older men, and 5) to test whether sleep disorders are associated with bone density and fracture risk in older men. The bank of MrOS specimens will be supplemented to allow for testing of future hypotheses concerning the role of sleep in the development of age-related diseases and conditions.

ELIGIBILITY:
No eligibility criteria

Ages: 65 Years to 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Older Adult
Dates: Start 2003-09; Primary Completion 2007-06 (Actual); Study Completion 2007-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Barrett-Connor — University of California, San Diego; Jane Cauley — University of Pittsburgh; Kristine Ensrud — University of Minnesota; Cora Lewis — University of Alabama at Birmingham; Eric Orwoll — Oregon Health and Science University; Susan Redline — Case Western Reserve University; Marcia Stefanick — Stanford University; Katie Stone — University of California, San Francisco

REFERENCES:
- [Derived] Hartmann S, Parrino L, Ensrud K, Stone KL, Redline S, Clark SR, Baumert M. Association between psychotropic medication and sleep microstructure: evidence from large population studies. J Clin Sleep Med. 2023 Mar 1;19(3):581-589. doi: 10.5664/jcsm.10394. PMID 36546402
- [Derived] Shahrbabaki SS, Linz D, Redline S, Stone K, Ensrud K, Baumert M. Sleep Arousal-Related Ventricular Repolarization Lability Is Associated With Cardiovascular Mortality in Older Community-Dwelling Men. Chest. 2023 Feb;163(2):419-432. doi: 10.1016/j.chest.2022.09.043. Epub 2022 Oct 13. PMID 36244405
- [Derived] May AM, May RD, Bena J, Wang L, Monahan K, Stone KL, Barrett-Connor E, Koo BB, Winkelman JW, Redline S, Mittleman MA, Mehra R; Osteoporotic Fractures in Men (MrOS) Study Group. Individual periodic limb movements with arousal are temporally associated with nonsustained ventricular tachycardia: a case-crossover analysis. Sleep. 2019 Oct 21;42(11):zsz165. doi: 10.1093/sleep/zsz165. PMID 31585012
- [Derived] Baumert M, Immanuel SA, Stone KL, Litwack Harrison S, Redline S, Mariani S, Sanders P, McEvoy RD, Linz D. Composition of nocturnal hypoxaemic burden and its prognostic value for cardiovascular mortality in older community-dwelling men. Eur Heart J. 2020 Jan 21;41(4):533-541. doi: 10.1093/eurheartj/ehy838. PMID 30590586